CLINICAL TRIAL: NCT04214340
Title: Current Management of Appendicitis in Adults and Children in France-A Prospective Study by the French Surgical Association Multicenter Cohort (APPEA)
Brief Title: Appendicitis in Adults and Children in France-A Prospective Study by the French Surgical Association Multicenter Cohort
Acronym: APPEA
Status: Completed | Type: Observational
Sponsor: Association Francaise de Chirurgie (Other)
Responsible Party: Principal Investigator, Pr Catherine Arvieux, Professor, Association Francaise de Chirurgie
Other Study IDs: AFC
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Appendicitis Acute; Peritonitis
Keywords: laparoscopic surgery
MeSH Terms: conditions — Appendicitis; Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: evaluation of practices — Study of the management and follow-up of patients presenting with appendicitis in France.

SUMMARY:
Acute appendicitis still represents a surgical challenge, despite profound changes in practice in recent decades. The objective of this study was comprehensively document current surgical practices aimed at improving the management and follow-up of pediatrics and adults patients presenting with appendicitis in France.

DETAILED DESCRIPTION:
The APPEA series is a national multicentric prospective cohort that included children and adults in France with acute appendicitis presenting between March 1st and June 30th, 2016. Data included demographic characteristics, medical history, symptoms, biology, radiology, treatments given during hospitalization, the modalities of the intervention, and any complications during a follow-up period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for appendicitis in participating centers
* informed

Exclusion Criteria:

* patient's (or parent's for children) opposition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admited in participating centers for acute appendicitis between 2016/03/01 and 2016/06/30
Sampling Method: Non-Probability Sample
Enrollment: 2285 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Surgical practices in the management of adults and pediatrics patients with appendicitis | 6 months
  Rate of laparoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: catherine ARVIEUX, MD, PHD, Principal Investigator — CHU Grenoble Alpes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhangu A, Soreide K, Di Saverio S, Assarsson JH, Drake FT. Acute appendicitis: modern understanding of pathogenesis, diagnosis, and management. Lancet. 2015 Sep 26;386(10000):1278-1287. doi: 10.1016/S0140-6736(15)00275-5. PMID 26460662
- [Background] Mak GZ, Loeff DS. Paradigm Shifts in the Treatment of Appendicitis. Pediatr Ann. 2016 Jul 1;45(7):e235-40. doi: 10.3928/00904481-20160525-01. PMID 27403670
- [Background] Teixeira FJR Jr, Couto Netto SDD, Akaishi EH, Utiyama EM, Menegozzo CAM, Rocha MC. Acute appendicitis, inflammatory appendiceal mass and the risk of a hidden malignant tumor: a systematic review of the literature. World J Emerg Surg. 2017 Mar 9;12:12. doi: 10.1186/s13017-017-0122-9. eCollection 2017. PMID 28286544
- [Background] Wagner M, Tubre DJ, Asensio JA. Evolution and Current Trends in the Management of Acute Appendicitis. Surg Clin North Am. 2018 Oct;98(5):1005-1023. doi: 10.1016/j.suc.2018.05.006. Epub 2018 Jul 13. PMID 30243444